CLINICAL TRIAL: NCT01112254
Title: Evaluation of the Diagnostic Performance of MRI±Biopsy to Optimize Resection of Ductal Carcinoma In Situ (DCIS) Breast Cancer
Acronym: IRCIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGR IRCIS 1503
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Ductal Carcinoma In Situ (DCIS) breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

ARMS (2):
- MRI±biopsy (Experimental): a MRI-guided or CT-guided preoperative biopsy will be performed in case of suspicious enhancement, multiple and large lesions (more than 3 cm from the initial lesion), not viewed on the mammography or breast ultrasound. The surgery type will depends on the MRI ± biopsy results.
  Interventions: Procedure: MRI±biopsy
- Standard care (No Intervention): The patients will be operated without additional exams

INTERVENTIONS:
Procedure: MRI±biopsy — A MRI-guided or CT-guided preoperative biopsy will be performed in case of suspicious enhancement, multiple and large lesions (more than 3 cm for from the initial lesion), which is not viewed on the mammography or breast ultrasound. The surgery type will depends on the MRI +/- ± biopsy results.
  Arms: MRI±biopsy

SUMMARY:
The purpose of this study is to evaluate the diagnostic performance of MRI±biopsy to optimize resection of Ductal Carcinoma In Situ (DCIS) breast cancer.

DETAILED DESCRIPTION:
Ductal carcinoma in situ (DCIS) is a frequent disease, concerning more than 15% of all breast carcinomas in France. Frequency increases due to breast screening programs. Breast conservative treatment can be done for limited lesions. Complete pathological excision with safe surgical margins is the main factor of success rate for conservative treatment. But safe surgical margins are not always obtained in the first surgery because preoperative or peroperative evaluation of the extent of the lesions is difficult. A 20 to 38% rate of involved margins is reported in the literature, implying a second surgery. MRI is not commonly performed today in the preoperative staging of DCIS, despite interesting results of breast MRI in DCIS evaluation published recently in a German study (Kuhl, Lancet 2007). Nevertheless, this retrospective study focused on a population of high-risk women (BRCA1-2 mutation carriers, family history of breast cancer…).

Additional suspicious lesions detected by MRI require MRI-guided or CT-guided biopsy as they are not detectable with mammography or ultrasound. Moreover, intraoperative pathological analysis cannot be performed in DCIS and surgical strategy will be different for a unique lesion (lumpectomy) or multiple/large lesions (mastectomy). If surgery is adapted according to MRI and biopsy results, we can assume that the entire lesion could be removed in a single operation, avoiding re-excisions, anxiety and reducing the costs.

The main objective of this protocol is to evaluate the value of MRI+biopsy in the staging of mammography-detected DCIS in an unselected population of women. It is a multicentric, randomised study including patients from France presenting a unique, limited (< 30 mm) DCIS detected by mammography or breast ultrasound. The two compared arms are: preoperative breast MRI+biopsy versus no additional diagnostic examination. High resolution dynamic 3D images will be obtained in order to detect very small suspicious lesions, typical of DCIS. The main endpoint is the re-excision rate for involved margins. In order to show a reduction of 50% of the rate of second surgery (from 25% to 12.5% in the MRI arm), it is necessary to include 360 patients (bilateral test, alpha=5%, power=80%).

A cost-effective study will be performed. The costs likely to differ between the two arms (MRI, biopsy, outpatient visits, hospitalisations, transportation, and sick leaves) will be assessed using data collected in the trial. The endpoint of the cost-effectiveness study will be the cost by success (cost-effectiveness ratio). A success is defined as achieving margin-negative resection after initial surgery (no need for re-excision). The other secondary endpoints will be to determine the rate of initial mastectomy and to describe MRI morphologic features in the MRI+biopsy arm.

ELIGIBILITY:
Inclusion Criteria:

* T0 or T1 breast DCIS revealed by microcalcifications on mammography + breast ultrasound
* Histological confirmation by percutaneous biopsy : strict DCIS or micro-invasive.
* Radiological focus < 30mm and accessible to conservative treatment.
* Single microcalcification focus
* Age : 18 to 80 years old
* Performance Status < 2
* Patient information and signed informed consent.

Exclusion Criteria:

* Invasive carcinoma
* Non biopsiable microcalcification focus under stereotaxy
* Bilateral lesions
* Non feasible MRI (claustrophobic, serious allergy, pace-maker, etc.)
* Refusal of surgery, including mastectomy if necessary
* History of homolateral breast cancer
* patient at risk of breast cancer (BRCA1 or 2 mutation or score 5 INSERM table)
* Pregnant or possibly pregnant or breastfeeding woman
* Person deprived of freedom or under guardianship
* Inability to undergo the medical surveillance of the trial for geographical, social or psychological reasons

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Re-excision rate | in the 6 months following randomization
  After histological confirmation of DCIS by stereotactic biopsy the patients will be randomized. In arm 1, a MRI-guided or CT-guided preoperative biopsy will be performed in case of suspicious enhancement, multiple and large lesions (more than 3 cm from the initial lesion), not viewed on the mammography or breast ultrasound. The surgery type will depends on the MRI ± biopsy results. The patients will be operated without additional exams in arm 2.

SECONDARY OUTCOMES:
Cost-effectiveness study | during the 6-month period after randomization
  cost by success, success being defined by the absence of re-excision during the 6-month period after randomization.
Relapse rate | at 30 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Balleyguier C, Dunant A, Ceugnart L, Kandel M, Chauvet MP, Cherel P, Mazouni C, Henrot P, Rauch P, Chopier J, Zilberman S, Doutriaux-Dumoulin I, Jaffre I, Jalaguier A, Houvenaeghel G, Guerin N, Callonnec F, Chapellier C, Raoust I, Mathieu MC, Rimareix F, Bonastre J, Garbay JR. Preoperative Breast Magnetic Resonance Imaging in Women With Local Ductal Carcinoma in Situ to Optimize Surgical Outcomes: Results From the Randomized Phase III Trial IRCIS. J Clin Oncol. 2019 Apr 10;37(11):885-892. doi: 10.1200/JCO.18.00595. Epub 2019 Feb 27. PMID 30811290
- See also: website of Institut Gustave Roussy — http://www.igr.fr/?p_lang=en